CLINICAL TRIAL: NCT04375189
Title: Impact of a Novel Complex Outpatient Clinic Setup on Patient Outcomes and Intern Education
Brief Title: High Risk Outpatient Intern-led Care (HeROIC) Clinic Initiative
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19, funding
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00137125
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Comorbidities and Coexisting Conditions; Risk Reduction; Emergencies
Keywords: High utilizer; High needs; Multimorbidity; Intensive outpatient care; Resident education
MeSH Terms: conditions — Risk Reduction Behavior; Emergencies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention)
- Complex Clinic Arm (Experimental)
  Interventions: Other: High Risk Clinic

INTERVENTIONS:
Other: High Risk Clinic — Subgroup of primary care clinic where patients have longer time slots, supervision by one longitudinal attending, "bedside" presentations
  Arms: Complex Clinic Arm

SUMMARY:
Background: A small subset of the patient population is responsible for a significant proportion of healthcare expenditures. These patients are cared for in academic medical centers by internal medicine residents however there has been no research to date about the education or the management of patients with complex multimorbidity in the outpatient setting.

Objective: To evaluate the impact of the High Risk Outpatient Intern-led Care (HeROIC) Clinic on internal medicine interns' perceived ability to manage complex outpatients as well as pre and post intervention total patient healthcare cost.

Methods: The investigators created the HeROIC outpatient clinic environment to comprise longer visit time slots, "bedside" presentations, and team-based care (one intern primary care provider, one secondary intern, and one longitudinal attending). All non-preliminary interns based at one primary care site participated in the intervention while interns at a second site continued to practice in the usual outpatient clinic environment. The interns in the HeROIC clinic arm assumed the roles of primary care providers for 34 complex patients in total. The primary outcome was the perceived confidence in the management of complex outpatients as assessed by a survey. Secondary outcomes included perceptions about the ability to provide high-quality outpatient and evidence-based outpatient care, as well as statewide pre-post patient healthcare cost data.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 6 medical comorbidities
* ≥ 2 admissions past 6 months or ≥ 4 past 1 year
* New or returning patient in resident primary care clinic

Exclusion Criteria:

* Primary mental health disease driving hospitalizations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Number of Inpatient or ER visits | Up to 2 years post enrollment
  Presentations to the ER and hospitalizations

SECONDARY OUTCOMES:
Total medical cost | Up to 2 years post enrollment
  Total medical costs (Outpatient, Inpatient, Imaging, Labs)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Epstein, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Outpatient Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No